CLINICAL TRIAL: NCT03524560
Title: Risk Factors for Polypharmacy in Older Adults in a Primary Care Setting:A Cross Sectional Study
Brief Title: Risk Factors for Polypharmacy in Older Adults
Status: Completed | Type: Observational
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, SULEYMAN ERSOY, Assist.Prof. Department of Family Medicine, Karabuk University
Other Study IDs: KBU-BAP-33/1-KA-077
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Polypharmacy
Keywords: comprehensive geriatric assesment, polypharmacy,geriatric depression scale,neutrophil/lymphocyte ratio

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Comprehensive geriatric assesment — Comprehensive Geriatric Assesment (CGA) consisting of detailed history and examination, drug consumption information, Body Mass Index (BMI), Waist Circumference (WC), Timed Up & Go test (TUG), Clock Drawing Test (CD), Activities of Daily Living and Instrumental Activities of Daily Living scales (ADL & IADL), Mini Mental State Examination (MMSE), Tinetti Gait and Tinetti Balance scores (TG &TB), 30 items Geriatric Depression Scale (GDS) was performed for each subject

SUMMARY:
Patients who were 65 years old or older and applied to Melek Hatun family practice center were enrolled in the study. All patients were seen either in our center or in their homes, and informed consents were obtained. Comprehensive Geriatric Assessment (CGA) was performed for each subject. Data were evaluated by PASW 17. The amount of medicines that the patient used everyday (DDC) was dependent variable. Relationships between DDC and other continuous variables were examined by Pearson's correlation. For categorical independent variables, t-tests were performed.

DETAILED DESCRIPTION:
1000 patients who were 65 years old or older and applied to Melek Hatun family practice center either in person or through a relative between 01 December 2014 and 01 August 2017 were enrolled in the study. All patients were seen either in our center or in their homes, and informed consents were obtained. Comprehensive Geriatric Assessment (CGA) consisting of detailed history and examination, drug consumption information, Body Mass Index (BMI), Waist Circumference (WC), Timed Up & Go test (TUG), Clock Drawing Test (CD), Activities of Daily Living and Instrumental Activities of Daily Living scales (ADL & IADL), Mini Mental State Examination (MMSE), Tinetti Gait and Tinetti Balance scores (TG &TB), 30 items Geriatric Depression Scale (GDS) was performed for each subject[8-16]. Additional tests like blood examinations or ECG were performed on the basis of necessity. Metabolic Syndrome (MS) was diagnosed according to WHO criteria [17].

Data were evaluated by PASW 17. The amount of medicines that the patient used everyday (Daily Drug Consumption-DDC) were dependent variable. Relationships between DDC and other continuous variables were examined by Pearson's correlation. For categorical independent variables, t-tests were performed. The variables which were found associated with DDC were controlled for confounding variables by linear regressions. To avoid collinearity problems, variables that were strongly interrelated (like CD and MMSE) were not added to the regression model together. For all analyses, the level of significance was assumed as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients of 65

Exclusion Criteria:

* Patients under 65 years
* Patients who do not want to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All of the patients who were 65 years old or older and applied to Melek Hatun family practice center either in person or through a relative between 01 December 2014 and 01 August 2017 were enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Daily drug consumption | 1 day
  Number of drugs used everyday

CONTACTS AND LOCATIONS:
Overall Officials: Selcuk Engin, Principal Investigator — Melekhatun family practice center

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the completion of the study data will be available
Access Criteria: among the colleagues who kindly request the data set by sending email to any of the authors will be given the url to reach the related data content
URL: https://goo.gl/wyq8QY